CLINICAL TRIAL: NCT05057026
Title: Impact of a Mental Health Support Program on Stigmatization and Confidence of Medical Residents Working With People With Mental Health Concerns
Brief Title: Impact of a Mental Health Support Program on of Medical Residents' Stigmatization Towards People With Lived Experience
Status: Terminated | Type: Observational
Why Stopped: Substantial efforts to engage participants in the evaluations was unsuccessful.
Sponsor: Bianca Horner (Other)
Collaborators: University of Calgary (Other)
Responsible Party: Sponsor-Investigator, Bianca Horner, Psychiatrist, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Other Study IDs: Version1, July 29, 2021
Record Dates: First submitted 2021-09-10; First posted 2021-09-27 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Depression, Anxiety Disorders
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult mental health support program: The investigators will evaluate the Impact of an Adult mental health support program on stigmatization and confidence of medical residents working with people with mental health concerns. The intervention will be delivered to approximately 30 residents from the University of Dalhousie family medicine residency program from the 2021-2022 academic year. The training will be delivered by resident groups. The first group will receive the PSP training October - November 2022. The second will receive the training November 2021 to February 2022. The third will take the training March to May 2022. Each group will include approximately 10 residents.
  Interventions: Other: Training Program Adult Mental Health Practice Support Program

INTERVENTIONS:
Other: Training Program Adult Mental Health Practice Support Program — The Adult Mental Health Practice Support Program (PSP) was designed in 2009 by the General Practice Services Committee (GPSC) to address needs expressed by the province's family physicians to improve patient care in British Colombia. Its content and delivery model has been designed using evidence-based key ingredients and implication factors understood to be important for effective stigma reduction. These include the following:
  * the use of contact-based education,
  * skills-building to increase confidence and provide another management option with or without drugs particularly if access to mental health support services is difficult or absent
  * tools - using the principles of cognitive behavioural theory
  The training will be delivered virtually over a total of 4 sessions two weeks apart, covering an 8-week period. A two hour virtually delivered booster session will be provided to students approximately one year after the delivery of the initial training.

SUMMARY:
The program, called the Mental Health Practice Support Program, is designed to teach new tools and skills for working with patients with mental health concerns in a family practice setting. The program is also being evaluated for effectiveness.

DETAILED DESCRIPTION:
Description of the Intervention

The Adult Mental Health Practice Support Program (PSP) was designed in 2009 by the General Practice Services Committee (GPSC) (a joint initiative of the BC Medical Association and the BC Ministry of Health) to address needs expressed by the province's family physicians to improve patient care in British Colombia. Its content and delivery model has been designed using evidence-based key ingredients and implication factors understood to be important for effective stigma reduction. These include the following:

* the use of contact-based education, a well-established best practice to reduce stigma where patients share their story with a focus on recovery, showing that recovery is not only possible but the goal;
* skills-building to increase confidence and provide another management option with or without drugs particularly if access to mental health support services is difficult or absent;
* tools - using the principles of cognitive behavioural theory -- than can be flexibly used within constraints of a busy practice reflecting a "real world" scenario;
* provider-patient shared responsibility in decision-making, patient engagement in recovery process
* practical practice support throughout the training period. The AMHPSP program has been implemented and evaluated with practicing primary care practitioners in numerous jurisdictions with positive results.

The program introduces learners to an organized approach to mental health treatment, starting from a problem and strength-based assessment through to the development of an action plan, which, using flow charts, providers can negotiate user-friendly CBT-based self-management options tailored to patient needs. These tools can be delivered within office time constraints, reflecting a "real world" scenario. One of the many tools is the AMHPSP algorithm, which houses all program tools and can be saved on a desktop for easy access at the click of a button (e.g., several validated screening scales for mental illnesses commonly seen in primary care, perinatal screening tools, medication algorithm, useful referral forms etc.) in addition to the three main supported self-management strategies described below:

* The Cognitive Behavioral Interpersonal Skills workbook (CBIS) The CBIS manual includes three main assessment tools: 1) the Diagnostic Assessment Interview; 2) the Problem List, Problem List Action Plan, and Resource list; and 3) the SAQ self-assessment questionnaires, all of which engage patient participation.
* The BounceBack program led by the Canadian Mental Health Association consists of a telephone delivered provincially funded evidence-based skills program designed to help adults experiencing symptoms of mild to moderate depression, low mood, or stress, with or without anxiety. Mental health coaches will work with patients usually every 1-2 weeks. The service operates at arm's length of HCPs all the while sending providers essential information on diagnosis and care course trajectory.

The primary thrust of the program is that all tools are meant to help build a shared responsibility model with the patient by increasing patient-provider interaction, negotiation, and partnership. Patients are encouraged to take an active role in the management of the problems most relevant to them, which in the end engages them in their recovery effort.

While previous implementations of the PSP program were delivered in-person, the adapted version for medical residents will be delivered virtually, to accommodate for any additional possible disruptions that may be brought about the ongoing COVID-10 pandemic.

Research Question and Objectives

The objective of the research is to assess the extent to which the adapted PSP program is effective at increasing residents' confidence and comfort in working with patients with mental health concerns; and decreasing stigmatizing attitudes, including the preference for social distance. Specific research questions are as follows:

The investigators hypothesize that enhanced skills in program participants will lead to increased comfort on the part of the medical residents, diminished preference for social distance, and improved attitudes and emotional responses towards patients with mental illnesses.

Methods The research is an intervention study, using a longitudinal pre-post-follow up design.

The intervention will be delivered virtually over a total of 4 sessions, covering an 8-week period. Each training session will take place approximately two weeks apart and will be two hours in length. A Practice Support Coordinator will support the "action period" work of the residents in between each of the training sessions. A two hour virtually delivered booster session will be provided to students approximately one year after the delivery of the initial training.

Outcomes of Interest

The investigators have identified two primary outcomes, which are as follows:

* Reduction in stigmatizing attitudes and behaviors from pre to post intervention, including preference for social distance, attitudes, and emotional responses toward patients with a mental illness.
* Improvements in confidence and comfort working with patients with mental health concerns from pre to post intervention.

Secondary outcomes are:

* Confidence and comfort in the use of tools/strategies.
* Impact of the program on emotional responses to interactions with patients with mental illnesses.

Our exploratory outcome of interest is an examination of the correlation between changes in stigma and changes in comfort or confidence.

The investigators will examine changes in mean scores across the different time points, using paired t-tests. A clinically meaningful outcome is considered as an improvement of 10% on the OMS-HC from pre to post training, which is slightly higher than the score change observed in a previous large scale RCT study of the PSP program with practicing physicians in Nova Scotia. Our calculations indicate that a sample of 26 residents will be required. Under this assumption, 80% power would be achieved to detect this difference with an alpha value of 5%.

A report on the results of the study will be compiled, with the intention that findings are publishable in the peer reviewed literature. Study findings will also be presented at academic conferences.

ELIGIBILITY:
Inclusion Criteria:

* Family Medicine residency program students in the1st year of their program.
* Provision of informed consent In good standing in their program.

Exclusion Criteria:

• Medical Students who are not enrolled in Dalhousie University Family Medicine residency program

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Residents from the University of Dalhousie family medicine residency program providing care for people with mental health conditions
Sampling Method: Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2021-10-05 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2022-06-10 (Actual)

PRIMARY OUTCOMES:
Opening Minds Scale for Health Providers (OMS-HC) | Pre-training, post-training, 6 , 12 and 18 months post -training
  Stigma changes will be measured using the 15 item Opening Minds Scale for Health Providers (OMS-HC), which captures providers' overall mental health related stigma as well as three main dimensions of stigma: negative attitudes, health professionals' own willingness to disclose/seek help for a mental illness, and preference for greater social distance. Total scores can range from 15 to 75, with lower scores indicating less stigma. This scale has been widely validated and used in evaluations of anti-stigma interventions in Canada. In 2014, a rigorous examination of the psychometric properties and responsiveness of the OMS-HC scale was conducted by Modgill G, et al. Results from this evaluation showed internal consistency as acceptable for all versions of the OMS scale (α = 0.74 to 0.79) and corresponding subscales (α = 0.67 to 0.68), further depicting the OMS-HC as an accurate and reliable instrument
PSP resident study_survey v1F Comfort in Managing Mental Health Conditions | Pre-training, post-training, 6 , 12 and 18 months post -training
  Confidence in managing depression will be assessed using adaptations of measures used in previous evaluations of this program with practicing primary care physicians. Modified versions of three ad hoc scales developed for a randomized controlled evaluation study in Nova Scotia were used to collect demographic information. The scales were also used to assess levels of confidence on a number of statements pertaining to their ability to diagnose, treat, and otherwise manage patients' mental health concerns using a 7-point Likert scale (not at all, very low, low, moderate, high, very high), with higher scores indicating higher levels of confidence, comfort, and familiarity.

SECONDARY OUTCOMES:
Emotion Scale | Pre-training, post-training, 6 , 12 and 18 months post -training
  The Emotion scale stigma uses10 item Emotion Scale, which assesses perceived emotional responses to interactions with patients with mental illnesses. Participants are instructed to imagine contact with a person with mental illness and to then rate the intensity of 10 emotions participants would experience during this encounter. Nine-point Likert scales (ranging from 1 = weak to 9 = strong) were used to assess the intensity of ten emotions: compassion, interest, sadness, acceptance, anger, dislike, anxiety, aversion, distrust and indifference. The selection of emotions was based on the assumption that these emotions are frequently experienced during the encounter with mentally ill individuals.
PSP resident study_survey v1F Use of and Comfort in Use of Tools and Strategies of the Program | Pre-training, post-training, 6 , 12 and 18 months post -training
  A modified version of of three ad hoc scales developed for a randomized controlled trial in Nova Scotia, the "PSP resident study_survey v1F Use of and Comfort in Use of Tools and Strategies of the Program" measures the use and reported comfort in the use of tools/skills, assessed through a series of simple yes/no responses pertaining to if the physician uses the tool, and measure levels of familiarity, confidence and comfort with program specific tools and skills taught in the program using a 7-point Likert scale (not at all, very low, low, moderate, high, very high).

OTHER OUTCOMES:
Correlation between changes in Physician Confidence and Stigma Scores. | Pre-training, post-training, 6 , 12 and 18 months post -training
  Our exploratory outcome is an examination of the correlation between changes in stigma and changes in comfort or confidence which will be assessed through regression analysis

CONTACTS AND LOCATIONS:
Overall Officials: Bianca Lauria-Horner, MD, Principal Investigator — Dalhousie University Department of Psychiatry
Locations (1):
- Dalhousie University Department of Psychiatry, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: Yes
Publication Conferences
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 36 Months

REFERENCES:
- [Result] Adshead, Gwen. 2005. Healing ourselves: ethical issues in the care of sick doctors. Advances in Psychiatric Treatment 11 (5): 330-37. https://doi.org/10.1192/apt.11.5.330.
- [Result] Azrin ST. Integrated care: High-impact mental health-primary care research for patients with multiple comorbidities. Psychiatr Serv. 2014 Apr 1;65(4):406-9. doi: 10.1176/appi.ps.201300537. PMID 24534819
- [Result] Beaulieu T, Patten S, Knaak S, Weinerman R, Campbell H, Lauria-Horner B. Impact of Skill-Based Approaches in Reducing Stigma in Primary Care Physicians: Results from a Double-Blind, Parallel-Cluster, Randomized Controlled Trial. Can J Psychiatry. 2017 May;62(5):327-335. doi: 10.1177/0706743716686919. Epub 2017 Jan 17. PMID 28095259
- [Result] Caldwell TM, Jorm AF. Mental health nurses' beliefs about likely outcomes for people with schizophrenia or depression: a comparison with the public and other healthcare professionals. Aust N Z J Ment Health Nurs. 2001 Mar;10(1):42-54. doi: 10.1046/j.1440-0979.2001.00190.x. PMID 11421972
- [Result] Health Nursing 10 (1): 42-54. https://doi.org/10.1046/j.1440-0979.2001.00190.x. College of Family Physicians of Canada, Canadian Psychiatric Association, and Canadian Psychological Association. (2020). Integrating Mental Health Services in Primary Care. Ontario: College of Family Physicians of Canada, Canadian Psychiatric Association, and Canadian Psychological Association.
- [Result] Corrigan P. How stigma interferes with mental health care. Am Psychol. 2004 Oct;59(7):614-625. doi: 10.1037/0003-066X.59.7.614. PMID 15491256
- [Result] Emrich K, Thompson TC, Moore G. Positive attitude. An essential element for effective care of people with mental illnesses. J Psychosoc Nurs Ment Health Serv. 2003 May;41(5):18-25. doi: 10.3928/0279-3695-20030501-09. PMID 12743963
- [Result] Jones S, Howard L, Thornicroft G. 'Diagnostic overshadowing': worse physical health care for people with mental illness. Acta Psychiatr Scand. 2008 Sep;118(3):169-71. doi: 10.1111/j.1600-0447.2008.01211.x. No abstract available. PMID 18699951
- [Result] Knaak S, Mantler E, Szeto A. Mental illness-related stigma in healthcare: Barriers to access and care and evidence-based solutions. Healthc Manage Forum. 2017 Mar;30(2):111-116. doi: 10.1177/0840470416679413. Epub 2017 Feb 16. PMID 28929889
- [Result] Knaak S, Modgill G, Patten SB. Key ingredients of anti-stigma programs for health care providers: a data synthesis of evaluative studies. Can J Psychiatry. 2014 Oct;59(10 Suppl 1):S19-26. doi: 10.1177/070674371405901s06. PMID 25565698
- [Result] Knaak S, Patten S. A grounded theory model for reducing stigma in health professionals in Canada. Acta Psychiatr Scand. 2016 Aug;134 Suppl 446:53-62. doi: 10.1111/acps.12612. PMID 27426646
- [Result] Kopera M, Suszek H, Bonar E, Myszka M, Gmaj B, Ilgen M, Wojnar M. Evaluating Explicit and Implicit Stigma of Mental Illness in Mental Health Professionals and Medical Students. Community Ment Health J. 2015 Jul;51(5):628-34. doi: 10.1007/s10597-014-9796-6. Epub 2014 Dec 23. PMID 25535045
- [Result] Lauria-Horner B, Beaulieu T, Knaak S, Weinerman R, Campbell H, Patten S. Controlled trial of the impact of a BC adult mental health practice support program (AMHPSP) on primary health care professionals' management of depression. BMC Fam Pract. 2018 Nov 28;19(1):183. doi: 10.1186/s12875-018-0862-y. PMID 30486799
- [Result] Lukovic JA, Miletic V, Pekmezovic T, Trajkovic G, Ratkovic N, Aleksic D, Grgurevic A. Self-medication practices and risk factors for self-medication among medical students in Belgrade, Serbia. PLoS One. 2014 Dec 11;9(12):e114644. doi: 10.1371/journal.pone.0114644. eCollection 2014. PMID 25503967
- [Result] MacCarthy D, Weinerman R, Kallstrom L, Kadlec H, Hollander MJ, Patten S. Mental health practice and attitudes of family physicians can be changed! Perm J. 2013 Summer;17(3):14-7. doi: 10.7812/TPP/13-033. PMID 24355885
- [Result] Modgill G, Patten SB, Knaak S, Kassam A, Szeto AC. Opening Minds Stigma Scale for Health Care Providers (OMS-HC): examination of psychometric properties and responsiveness. BMC Psychiatry. 2014 Apr 23;14:120. doi: 10.1186/1471-244X-14-120. PMID 24758158
- [Result] Nyblade L, Stockton MA, Giger K, Bond V, Ekstrand ML, Lean RM, Mitchell EMH, Nelson RE, Sapag JC, Siraprapasiri T, Turan J, Wouters E. Stigma in health facilities: why it matters and how we can change it. BMC Med. 2019 Feb 15;17(1):25. doi: 10.1186/s12916-019-1256-2. PMID 30764806
- [Result] Patten SB, Remillard A, Phillips L, Modgill G, Szeto ACh, Kassam A, Gardner DM. Effectiveness of contact-based education for reducing mental illness-related stigma in pharmacy students. BMC Med Educ. 2012 Dec 5;12:120. doi: 10.1186/1472-6920-12-120. PMID 23216787
- [Result] Schwenk TL, Davis L, Wimsatt LA. Depression, stigma, and suicidal ideation in medical students. JAMA. 2010 Sep 15;304(11):1181-90. doi: 10.1001/jama.2010.1300. PMID 20841531
- [Result] Sullivan GM, Feinn R. Using Effect Size-or Why the P Value Is Not Enough. J Grad Med Educ. 2012 Sep;4(3):279-82. doi: 10.4300/JGME-D-12-00156.1. No abstract available. PMID 23997866
- [Result] Ungar T, Knaak S, Szeto AC. Theoretical and Practical Considerations for Combating Mental Illness Stigma in Health Care. Community Ment Health J. 2016 Apr;52(3):262-71. doi: 10.1007/s10597-015-9910-4. Epub 2015 Jul 15. PMID 26173403
- [Result] Wallace JE. Mental health and stigma in the medical profession. Health (London). 2012 Jan;16(1):3-18. doi: 10.1177/1363459310371080. Epub 2010 Dec 22. PMID 21177717
- [Result] Weinerman R, Campbell H, Miller M, Stretch J, Kallstrom L, Kadlec H, Hollander M. Improving mental healthcare by primary care physicians in British Columbia. Healthc Q. 2011;14(1):36-8. doi: 10.12927/hcq.2011.22146. PMID 21301237
- [Result] MacCarthy D, Kallstrom L, Kadlec H, Hollander M. Improving primary care in British Columbia, Canada: evaluation of a peer-to-peer continuing education program for family physicians. BMC Med Educ. 2012 Nov 9;12:110. doi: 10.1186/1472-6920-12-110. PMID 23140230